CLINICAL TRIAL: NCT04946383
Title: The Safety and Effectivness of Quercetin and Dasatinib on the Epigenetic Aging Rates in Healthy Individuals
Brief Title: Safety and Effectivness of Quercetin & Dasatinib on Epigenetic Aging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TruDiagnostic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHB-QD-001
Record Dates: First submitted 2021-06-11; First posted 2021-06-30 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Aging
Keywords: Quercetin; Dasatinib; Epigenomics
MeSH Terms: interventions — Dasatinib; Quercetin

STUDY DESIGN:
Intervention Model Description: prospective non-randomized clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quercetin and Dasatinib supplements (Experimental): 500mg Quercetin and 50mg Dasatinib oral capsules on Monday, Tuesday, Wednesday (3 days in a row) per month for the duration of 6 months.
  Interventions: Drug: Dasatinib plus Quercetin

INTERVENTIONS:
Drug: Dasatinib plus Quercetin — Dasatinib plus Quercetin

SUMMARY:
Assessing the effects of Quercitin and Dasatinib over a 16 week period on participatns' epigenetic biological aging. The patients are being tested at baseline, halfway point, and after the trial period.

DETAILED DESCRIPTION:
This is a prospective non-randomized clinical study of 20-25 patients to evaluate the effectiveness of Quercetin and Dasatinib supplements on the patient's epigenetic aging rate. The investigators predict that Quercetin and Dasatinib combined will slow cell proliferation and thus decelerate the rate of aging.

There is evidence that Quercetin and Dasatinib slows cell proliferation and decelerates aging and the risk of age-related diseases. The aim of this pilot study is to evaluate the safety, efficacy and feasibility of Quercetin and Dasatinib as an effective treatment option to improve clinical care of healthy individual's epigenetic aging rate thus prolonging longevity.

Despite considerable effort, successful treatment of reversing one's biological age has been shown to be a difficult therapeutic challenge. There is evidence that Dasatinib+Quercetin(Quercetin and Dasatinib) is a safe and effective treatment option to improve clinical care of healthy individual's biological age. Studies have shown that Dasatinib+Quercetin slows cell proliferation and decelerates aging and the risk of age-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Ages 40 and older
* Patient must be able to comply with treatment plan and laboratory tests

Exclusion Criteria:

* Neoplastic cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
* No immune system issues or immunodeficiency disease
* No history of viral illness which could be reactivated by immune down regulation
* Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke)
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Patients infected with hepatitis, C or HIV
* Patients with Body Mass Index (BMI) > 40 kg/m2
* Presence of active infection 9. Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the investigator would render a patient unsuitable to participate in the study
* Unable or unwilling to provide required blood sample for testing
* As for the male-participants they are recommended to avoid fertilization for the first 6 months after the clinical trial.
* If the patient has previously used Quercetin and Dasatinib.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age Test | Change from baseline to 6 months

SECONDARY OUTCOMES:
Examining Methylation changes | Change from baseline to 6 months
  Methylation analysis via the Illumina 850k epic array. Methylation will be assessed at 850,000 spots on the DNA, these are located on CpG sites. These are the spots on DNA that have cytosine and guanine right next to each other.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Lee, MD, Principal Investigator — The Institute for Hormonal Balance
Locations (1):
- The Institute for Hormonal Balance, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavalcante MB, Saccon TD, Nunes ADC, Kirkland JL, Tchkonia T, Schneider A, Masternak MM. Dasatinib plus quercetin prevents uterine age-related dysfunction and fibrosis in mice. Aging (Albany NY). 2020 Jan 18;12(3):2711-2722. doi: 10.18632/aging.102772. Epub 2020 Jan 18. PMID 31955151
- [Background] Hickson LJ, Langhi Prata LGP, Bobart SA, Evans TK, Giorgadze N, Hashmi SK, Herrmann SM, Jensen MD, Jia Q, Jordan KL, Kellogg TA, Khosla S, Koerber DM, Lagnado AB, Lawson DK, LeBrasseur NK, Lerman LO, McDonald KM, McKenzie TJ, Passos JF, Pignolo RJ, Pirtskhalava T, Saadiq IM, Schaefer KK, Textor SC, Victorelli SG, Volkman TL, Xue A, Wentworth MA, Wissler Gerdes EO, Zhu Y, Tchkonia T, Kirkland JL. Senolytics decrease senescent cells in humans: Preliminary report from a clinical trial of Dasatinib plus Quercetin in individuals with diabetic kidney disease. EBioMedicine. 2019 Sep;47:446-456. doi: 10.1016/j.ebiom.2019.08.069. Epub 2019 Sep 18. PMID 31542391
- [Background] Ermogenous C, Green C, Jackson T, Ferguson M, Lord JM. Treating age-related multimorbidity: the drug discovery challenge. Drug Discov Today. 2020 Aug;25(8):1403-1415. doi: 10.1016/j.drudis.2020.06.016. Epub 2020 Jun 20. PMID 32574698